CLINICAL TRIAL: NCT00971646
Title: Cohort Study: Perceptual Urge Sensation
Status: Completed | Type: Observational
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 09-1234567
Record Dates: First submitted 2009-09-03; First posted 2009-09-04 (Estimated); Last update posted 2018-09-06 (Actual); Status verified 2018-09

CONDITIONS: Urinary Bladder, Overactive; Osteoporosis
Keywords: overactive bladder; self-consciousness; perceptual urge sensation
MeSH Terms: conditions — Urinary Bladder, Overactive; Osteoporosis | interventions — 4-amino-4'-hydroxylaminodiphenylsulfone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- OAB: Patients with overactive bladder syndrome
  Interventions: Other: Micturition diary; Other: Hospital Anxiety and Depression scale; Other: EuroQol-5D; Other: Self-consciousness questionnaire
- Osteoporosis: Patients with osteoporosis
  Interventions: Other: Micturition diary; Other: Hospital Anxiety and Depression scale; Other: EuroQol-5D; Other: Self-consciousness questionnaire

INTERVENTIONS:
Other: Micturition diary — On the micturition diary patients are asked to note every void and drink. With every void they are asked to estimate their bladder volume and grade their degree of desire to void.
Other: Hospital Anxiety and Depression scale — This questionnaire is designed to screen for the presence of a mood disorder.
Other: EuroQol-5D — This questionnaire grades the health condition of the subject.
Other: Self-consciousness questionnaire — The questions tap cognitive, emotional, and physical appearance aspects of directing their attention to the self.

SUMMARY:
Over the past few years it has become clear that our understanding of bladder physiology is inadequate to explain urge incontinence. This has forced us to re-evaluate what we know and do not know about bladder function and dysfunction. This has led to the identification and study of novel systems within the bladder that may contribute to abnormal sensations.

The investigators now suspect that the organic changes occurring in the bladder are not the whole story. For one group of patients with pathological urge there is growing evidence suggesting that there may be a strong psychological component. The idea now being put forward is that normal afferent peripheral information is perceived as abnormal and excessive, resulting in an increased desire to go to the bathroom: 'perceptual urge'. It is important to identify this group of patients since it will direct their treatment towards more cognitive approaches. Also, if such a psychological aetiology can be eliminated it would lead to a more focused and effective management of peripheral pathology with surgery or pharmacology.

ELIGIBILITY:
Inclusion Criteria (for patients with OAB):

* Patients older than 18 years with OAB diagnosed by their urologist using the criteria of more than 8 micturitions on three consecutive days of these three days they keep a micturation diary with a VAS score for urge sensation.

Patients should have at least one episode of urge: sudden compelling desire to void which can not be postponed.

* Well versed in Dutch.

Inclusion Criteria (for patients with osteoporosis):

* Patients older than 18 years with osteoporosis joined into the Fast Guide cohort program.
* Well versed in Dutch.

Exclusion Criteria (for patients with OAB):

* Patients with stress-urinary incontinence
* Presence of post void residual urine > 100cc determined by ultrasound
* Presence of urinary tract infection, determined by urine sticks. Patients with urinary tract infection will be treated by antibiotics. After resolution of the infection, the patient can re-enter the study if the urine is sterile at that moment.

Exclusion Criteria (for patients with osteoporosis):

* Urinary complaints or urologic history
* Presence of postvoid residual urine > 100cc determined by ultrasound
* Presence of urinary tract infection, determined by urine sticks. Patients that present with urinary tract infection will be definitively excluded from participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of two groups: 1: patients with OAB; 2: patients with osteoporosis.
  The patients with OAB will be reqruited from the outpatient clinic and website designed for patients with overactive bladder symptoms.
  The patients with osteoporosis will be recruited from an electronic patient database.
Sampling Method: Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2010-06 (Actual); Primary Completion 2017-03-01 (Actual); Study Completion 2017-03-01 (Actual)

PRIMARY OUTCOMES:
Defining differences in self-consciousness and HADS scores in patients with OAB | 1 year

SECONDARY OUTCOMES:
Defining differences between self-consciousness and HADS scores between the two cohorts | 1 year
Defining differences in quality of life between the two cohorts | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Gommert van Koeveringe, MD, PhD, urologist, Study Director — Maastricht University Medical Centre
Locations (1):
- Maastricht University Medical Centre, Maastricht, Limburg, Netherlands